CLINICAL TRIAL: NCT04071990
Title: Impact of Involvement of the Family in the Cognitive Behavioral Group Therapy for Obsessive-Compulsive Disorder: a Randomized Controlled Trial.
Brief Title: Family Involvement in CBGT of OCD: a Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BC-5080
Record Dates: First submitted 2019-08-02; First posted 2019-08-28 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Family based intervention; Cognitive behavioral group therapy; Exposure and response prevention; Family accommodation
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Intervention Model Description: After randomization the patient an family member will be allocated to one of the two groups: (a) CBGT with involvement of family (intervention) or (b) CBGT without involvement of family (control), both groups will exist of 12 sessions
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Family-based cognitive behavioral group therapy (FB-CBGT) (Active Comparator): One family member of each patient will be involved during all 12 CBGT sessions. The CBGT program that will be employed in the present study is a protocoled therapy consisting of psychoeducation, ERP techniques, cognitive tools to change dysfunctional thoughts and beliefs, strategies to prevent relapses, discussion on the family involvement (e.g. FA, burden, …) and homework exercises after each session.
  Interventions: Behavioral: FB-CBGT
- Cognitive-behavioral group therapy (CBGT) without family (Placebo Comparator): Each patient will be involved during all 12 CBGT sessions. The CBGT program that will be employed in the present study is a protocoled therapy consisting of psychoeducation, ERP techniques, cognitive tools to change dysfunctional thoughts and beliefs, strategies to prevent relapses, discussion on the family involvement (e.g. FA, burden, …) and homework exercises after each session., without the involvement of family members.
  Interventions: Behavioral: CBGT

INTERVENTIONS:
Behavioral: FB-CBGT — CBGT for OCD patients, with Involvement of family members (partner, parent, sibling, ...)
  Arms: Family-based cognitive behavioral group therapy (FB-CBGT)
Behavioral: CBGT — CBGT for OCD patients, without involvement of family members
  Arms: Cognitive-behavioral group therapy (CBGT) without family

SUMMARY:
With a lifetime prevalence of 1-3% Obsessive-Compulsive Disorder (OCD) is a chronic and disabling psychiatric disorder with considerable burden for the individual and society. Cognitive-behavioural group therapy (CBGT) is effective in reducing the intensity of OCD symptoms and it improves the OCD patient's quality of life. There is also growing evidence that family accommodation (FA) maintains and/or facilitates OCD symptoms, reinforces fear and avoidance behaviours in patients with OCD and is associated with family burden. Considering the promising results of involvement of family in CBGT on OCD symptoms and FA, the current study aims at investigating the effects of the involvement of the family in a 12-week CBGT protocol on the OCD symptoms, FA, burden, QOL, anxiety and depressive symptoms in OCD patients and their live-in relatives. Eighty patients with OCD and their live-in family members (partner, parent, sibling, …) between 18-65 years old will be included in this randomized controlled trial. Patients and family members will be randomly assigned to CBGT with the involvement of family or to CBGT without involvement of family. The primary goal of this study is to evaluate the effects of the involvement of live-in family members during a 12-week CBGT on OCD symptomatology and family accommodation during a 12-month follow-up period. In a secondary stage, we will explore whether the involvement of live-in family members during a 12-week CBGT will ameliorate anxiety and depressive symptoms, QOL, family functioning and burden in the patients and their live-in family.

DETAILED DESCRIPTION:
Participants will be recruited at the Centre for OCD at the Ghent University Hospital (UZ Gent) located in Belgium. A group of 80 patients and 80 live-in family members (partner, parent, sibling), between 18 and 65 years old. The patients with OCD will be selected based on the Diagnostic and Statistical Manual (DSM-5) diagnostic criteria for obsessive-compulsive disorder using the semi-structured Mini International Neuropsychiatric Interview (MINI screening version 7.0.2)(60). Other inclusion criteria are (a) the OCD patient with a score of at least 16 on the Yale-Brown Obsessive Compulsive Scale (Y-BOCS), (b) patient and family member fluent in Dutch and (c) both willing to attend all treatment sessions together. To maximize the generalizability of our sample, we did not exclude patients if they had comorbid mood or anxiety disorders, as long as OCD was the principal diagnosis. Patients and family members will be recruited before randomization, because the aim of this study is to investigate the impact of the involvement of the family in the CBGT. At the start of the experiment we will ask patients and their family members to sign the informed consent. Randomization occurs after oral and written informed consent and patients and family members will be notified about the treatment condition after randomization. After randomization the patient and family member will be allocated to one of the two treatment arms: (a) CBGT with involvement of family of family-based CBGT (FB-CBGT) (intervention) or (b) CBGT without involvement of family (control). The CBGT program exists of a fixed 12-week protocol, involving psycho-education, exposure and response prevention (ERP), cognitive restructuring, and the discussion about the family system.

ELIGIBILITY:
Inclusion Criteria:

* the OCD patient with a score of at least 16 on Y-BOCS
* patient and family member fluent in Dutch
* patient and family member both willing to attend all treatment sessions together.

Exclusion Criteria:

* current severe suicidality
* current substance abuse
* psychotic symptoms and
* OCD treated with deep brain stimulation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-09-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Faster decrease and longer lasting improvement (less relapse) of OCD symptoms in patients | Y-BOCS will be completed at four time-points: at inclusion, after completion of the CBGT (an average of 3 months post baseline) and at 6 and 12 months post CBGT
  Improvement of OCD symptoms will be measured by the Y-BOCS
Faster decrease and longer lasting improvement of family accommodation in family members | The Family Accommodation Scale (FAS) will be completed at four time-points: at inclusion, after completion of the CBGT (an average of 3 months post baseline) and at 6 and 12 months post CBGT
  Improvement of family accommodation will be measured by the family accommodation scale (FAS)

SECONDARY OUTCOMES:
A reduction in anxiety and depression in patients and family members | The HADS will be completed at four time-points: at inclusion, after completion of the CBGT (an average of 3 months post baseline) and at 6 and 12 months post CBGT
  The Hospital Anxiety and Depressive Scale (HADS) will be used to measure the presence of depression and anxiety and changes in depression and anxiety rates
Increase of quality of life (QOL) in patients | The WHOQOL-BREF will be completed at four time-points: at inclusion, after completion of the CBGT (an average of 3 months post baseline) and at 6 and 12 months post CBGT
  The Quality of Life Questionnaire (WHOQOL-BREF) will be administered to assess the perceived quality of life and emotional well-being in patients
An improvement in family functioning measured by the SCORE-15 in patients and family members | The SCORE-15 will be completed at four time-points: at inclusion, after completion of the CBGT(an average of 3 months post baseline) and at 6 and 12 months post CBGT
  The Systemic Clinical Outcome and Routine Evaluation 15-item version (SCORE-15) will be administered to assess the outcome in systemic family therapy and other family-oriented services
An improvement in family functioning measured by the BPNSFS in patients and family members | The BPNSFS will be completed at four time-points: at inclusion, after completion of the CBGT (an average of 3 months post baseline) and at 6 and 12 months post CBGT
  The Basic Psychological Need Satisfaction and Frustration Scale (BPNSFS) -addresses both need satisfaction and frustration in relationships. Whereas need satisfaction is associated with well-being, need frustration is associated with ill-being. Self-determination theory posits three universal psychological needs: autonomy; competence; and relatedness, and suggests that these must be present satisfactorily for people to maintain optimal performance and well-being.
An improvement in family functioning measured by the perceived criticism measure (PCM) in patients and family members | The PCM will be completed at four time-points: at inclusion, after completion of the CBGT (an average of 3 months post baseline) and at 6 and 12 months post CBGT
  The perceived criticism measure (PCM) consists of a 10-point Likert-type scale to describe a relative's degree of criticism of him of her. The patients' perception on their relatives' behavior may be the proximal factor in expressed emotions relationship to treatment response and relapse. This measure proved to be a strong predictor of outcome for outpatients with OCD.
A decrease of burden in family members | The ZBI will be completed at four time-points: at inclusion, after completion of the CBGT (an average of 3 months post baseline) and at 6 and 12 months post CBGT
  Family burden will be evaluated with the Zarit Burden Interview (ZBI) 22-item version, a self-report measure. The ZBI assesses the perceived burden in the caregivers of patients with psychiatric disorders.
Evaluation therapeutic sessions | The SRS will be completed at 12 time-points: after all therapeutic sessions, 12 sessions in total, during 3 months
  In order to assess how patients and family members evaluate the therapeutic relation, goals and topics, approach during the therapeutic session the Session Rating Scale (SRS V.3.0) will be administered.

CONTACTS AND LOCATIONS:
Overall Officials: Gilbert MD Lemmens, MD, PhD, Principal Investigator — Ghent University Hospital, University Ghent; Kurt Audenaert, MD, PhD, Principal Investigator — Ghent University Hospital, University Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No
The datasets generated and/or analyzed during the current study are not publicly available due to confidentiality issues but are available from the corresponding author upon reasonable request.